CLINICAL TRIAL: NCT06449209
Title: A Phase II, Multi-site, Open-label, Parallel Group Trial of BNT327 in Combination With Chemotherapy for Participants With Untreated Extensive-stage Small-cell Lung Cancer and Participants With Previously Treated Small-cell Lung Cancer
Brief Title: Safety, Preliminary Effectiveness of BNT327, an Investigational Therapy for Patients With Small-cell Lung Cancer in Combination With Chemotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BNT327-01
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Extensive-stage Small-cell Lung Cancer; Small-cell Lung Cancer
Keywords: Programmed Death-1 (PD-1); Programmed Death Ligand-1 (PD-L1); Programmed Death-1 monoclonal antibodies; Combination chemotherapy; Anti vascular endothelial growth factor (VEGF); Previously treated small-cell lung cancer; Untreated extensive-stage small-cell lung cancer; Dose optimization; Time to progression
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Etoposide; Carboplatin; Paclitaxel; Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 Arm 1 - BNT327 DL1 + carboplatin + etoposide (Experimental): Participants with ES-SCLC without prior systemic anticancer therapy received in the ES setting
  Interventions: Drug: BNT327 Dose Level 1 (DL1); Drug: Etoposide; Drug: Carboplatin
- Cohort 1 Arm 2 - BNT327 DL2 + carboplatin + etoposide (Experimental): Participants with ES-SCLC without prior systemic anticancer therapy received in the ES setting
  Interventions: Drug: BNT327 Dose Level 2 (DL2); Drug: Etoposide; Drug: Carboplatin
- Cohort 2 Arm 1 - BNT327 DL1 + paclitaxel (Experimental): Participants with SCLC who have disease progression/relapse
  Interventions: Drug: BNT327 Dose Level 1 (DL1); Drug: Paclitaxel
- Cohort 2 Arm 2 - BNT327 DL2 + paclitaxel (Experimental): Participants with SCLC who have disease progression/relapse
  Interventions: Drug: BNT327 Dose Level 2 (DL2); Drug: Paclitaxel
- Cohort 3 Arm 1 - BNT327 DL1 + topotecan (Experimental): Participants with SCLC who have disease progression/relapse
  Interventions: Drug: BNT327 Dose Level 1 (DL1); Drug: Topotecan
- Cohort 3 Arm 2 - BNT327 DL2 + topotecan (Experimental): Participants with SCLC who have disease progression/relapse
  Interventions: Drug: BNT327 Dose Level 2 (DL2); Drug: Topotecan

INTERVENTIONS:
Drug: BNT327 Dose Level 1 (DL1) — Intravenous (IV) infusion
  Arms: Cohort 1 Arm 1 - BNT327 DL1 + carboplatin + etoposide; Cohort 2 Arm 1 - BNT327 DL1 + paclitaxel; Cohort 3 Arm 1 - BNT327 DL1 + topotecan
Drug: BNT327 Dose Level 2 (DL2) — IV infusion
  Arms: Cohort 1 Arm 2 - BNT327 DL2 + carboplatin + etoposide; Cohort 2 Arm 2 - BNT327 DL2 + paclitaxel; Cohort 3 Arm 2 - BNT327 DL2 + topotecan
Drug: Etoposide — IV infusion
  Arms: Cohort 1 Arm 1 - BNT327 DL1 + carboplatin + etoposide; Cohort 1 Arm 2 - BNT327 DL2 + carboplatin + etoposide
Drug: Carboplatin — IV infusion
  Arms: Cohort 1 Arm 1 - BNT327 DL1 + carboplatin + etoposide; Cohort 1 Arm 2 - BNT327 DL2 + carboplatin + etoposide
Drug: Paclitaxel — IV infusion
  Arms: Cohort 2 Arm 1 - BNT327 DL1 + paclitaxel; Cohort 2 Arm 2 - BNT327 DL2 + paclitaxel
Drug: Topotecan — IV infusion or oral capsules
  Arms: Cohort 3 Arm 1 - BNT327 DL1 + topotecan; Cohort 3 Arm 2 - BNT327 DL2 + topotecan

SUMMARY:
This is a Phase II, multi-site, open-label, parallel group study in participants with untreated extended-stage small-cell lung cancer (ES-SCLC) (Cohort 1) or small-cell lung cancer (SCLC) which has progressed on first- or second-line treatment (Cohort 2 and Cohort 3). This study will assess the safety, efficacy, and pharmacokinetics (PK) of BNT327.

DETAILED DESCRIPTION:
In Cohort 1 of this study, two dose levels of BNT327 will be studied in combination with etoposide and carboplatin to identify an optimized dose for future clinical investigation.

Cohort 2 and Cohort 3 will explore the combination of two dose levels of BNT327 with paclitaxel, or topotecan in the second- or third-line setting.

Patients will be treated until disease progression, intolerable toxicity, patient withdrawal, study termination or up to 2 years (whichever occurs first).

Participants will be assigned to either Cohort 1 or Cohort 2/Cohort 3 based on their disease type (i.e., untreated ES-SCLC for Cohort 1 and SCLC which has progressed on first- or second-line treatment for Cohort 2 and Cohort 3). Assignment to either Cohort 2 or Cohort 3 will be the investigator's choice.

Participants will be randomized to each arm within each cohort:

* Participants enrolled to Cohort 1 and Cohort 3 will be randomized in a 1:1 ratio to Arm 1 or Arm 2.
* Participants enrolled to Cohort 2 will be randomized in a 2:1 ratio to Arm 1 or Arm 2.

ELIGIBILITY:
Inclusion Criteria (applicable to all participants unless otherwise specified):

* Cohort 1 only: Have histologically or cytologically confirmed ES-SCLC (using the American Joint Committee on Cancer [AJCC]) tumor node metastasis [TNM] staging system combined with Veterans Administration Lung Study Group two-stage classification scheme). For AJCC TNM staging system: AJCC 8th edition stage IV (T any, N any, M1a/b/c), or T3~4 for multiple lung nodules or tumor/nodule volume that cannot be encompassed in a tolerable radiotherapy plan.
* Cohort 1 only: Participants who have not received systemic therapy for ES-SCLC for various reasons including potential intolerance of the standard-of-care per the patient's treating physician's judgment. However, participants with prior chemoradiotherapy for Limited-Stage Small-Cell Lung Cancer (LS-SCLC) must have been treated with curative intent and had a treatment-free interval of at least 6 months since the last systemic anticancer treatment including chemotherapy, radiotherapy, or chemoradiotherapy before the diagnosis of ES-SCLC to be eligible.
* Cohort 2 and Cohort 3 only: Participants with SCLC who have disease progression/relapse after first-line platinum-based chemotherapy with or without immunotherapy, or after first-line platinum-based chemotherapy and one second-line of chemotherapy (not the same chemotherapy agent in the specific arm to be enrolled to) with time to progression ≥3 months during second-line treatment.
* Have given informed consent by signing and dating an informed consent form before initiation of any study-specific procedures.
* Male or female, aged ≥18 years at the time of giving informed consent.
* Are willing and able to comply with scheduled visits, treatment schedule, the planned study assessments, laboratory tests, lifestyle restrictions, and other requirements of the study. This includes that they are able to understand and follow study-related instructions.
* Have at least one measurable lesion as the targeted lesion based on RECIST 1.1. Lesions treated after prior local treatment (radiotherapy, ablation, interventional procedures, etc.) are generally not considered as target lesions. If the lesion with prior local treatment is the only targeted lesion, evidence-based radiology must be provided to demonstrate disease progression (the single bone metastasis or the single central nervous system metastasis should not be considered as a measurable lesion).
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Have a minimum life expectancy of >3 months.
* Have adequate organ function, as defined below:

  * Hematology:

    * Absolute neutrophil count ≥1.5 × 10^9/L.
    * Platelet count ≥100 × 10^9/L.
    * Hemoglobin ≥90 g/L or 5.6 mmol/L.
  * Liver function:

    * Total bilirubin ≤1.5 × upper limit of normal (ULN).
    * With Gilbert's syndrome total bilirubin <3 mg/dL and direct bilirubin ≤ULN. Note, Gilbert's syndrome must be documented appropriately as past medical history.
    * Participants without liver metastasis alanine aminotransferase and aspartate aminotransferase ≤2 × ULN.
    * Participants with liver metastasis alanine aminotransferase and aspartate aminotransferase ≤5 × ULN.
    * Albumin ≥3.0 g/dL.
  * Renal function: Serum creatinine ≤1.5 × ULN or creatinine clearance ≥50 mL/min. Cockcroft-Gault formula.
  * Qualitative urine protein ≤1+. If qualitative urine protein ≥2+, a 24-hour urine protein quantitative test is required. If the 24-hour urine protein result is <1 g, the participant can be enrolled.
  * Coagulation function: International normalized ratio or prothrombin time and activated partial thromboplastin time ≤1.5 × ULN unless the participant is receiving anticoagulation therapy as long as prothrombin or activated partial thromboplastin is within therapeutic range of intended use of anticoagulant.
* Are women of childbearing potential (WOCBP) who have a negative serum beta-human chorionic gonadotropin test at screening and before each IMP dose. Women born female that are postmenopausal (defined as 12 months with no menses without an alternative medical cause) or permanently sterilized (verified by medical records) will not be considered WOCBP and therefore will not be required to undergo pregnancy testing.
* Are WOCBP who agree to practice a highly effective form of contraception and to require their male sexual partners to use barrier contraception methods (preferably condoms), starting at Screening and continuously until 6 months after receiving the last study treatment.
* Are men who are sexually active with a partner born female and have not had a vasectomy who agree to use condoms and to ask their sexual partners to practice a highly effective form of contraception during the study, starting at the Screening Period and continuously until 6 months after receiving the last dose of IMP.
* Are WOCBP who agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study, starting at the Screening Period and continuously 6 months after receiving the last dose of IMP.
* Are men who are willing to refrain from sperm donation, starting at the Screening Period and continuously until 6 months after the last dose of IMP.

Exclusion Criteria (applicable to all participants):

* Are pregnant or breastfeeding or are planning pregnancy or planning to father children during the study or within 6 months after the last dose of IMP.
* Have a medical, psychological, or social condition which, in the opinion of the investigator, could compromise their wellbeing if they participate in the study, or that could prevent, limit, or confound the protocol-specified assessments or procedures, or that could impact adherence to protocol-described requirements.
* Have histologically or cytologically confirmed SCLC with combined histologies.
* Have received any of the following therapies or drugs within the noted time intervals prior to the initiation of study treatment:

  * Within 2 weeks: small molecule targeted agents with half-life of <7 days; or radiation not involving the thoracic cavity; local radiation for brain lesion is allowed; local radiation for bone lesions is allowed.
  * Within 4 weeks: radiation involving the thoracic cavity; small molecule targeted agents with half-life of ≥7 days; monoclonal antibodies, antibody-drug conjugates, radioimmunoconjugates, or T-cell or other cell-based therapies.
  * Participants who received prior treatment with a PDL-1/VEGF bispecific antibody.
  * Have received systemic corticosteroids (at a dosage greater than 10 mg/day of prednisone or an equivalent dose of other corticosteroids) within 10 days prior to the initiation of study treatment. Note: The following are allowed: local, intranasal, intraocular, intra-articular or inhaled corticosteroids, short-term use (≤7 days) of corticosteroids for prophylaxis (e.g., prevention of contrast agent allergy) or treatment of non-autoimmune conditions (e.g., delayed hypersensitivity reactions caused by exposure to allergens).
  * Have been vaccinated with live attenuated vaccine(s) within 4 weeks prior to initiation of the study treatment.
  * Received broad-spectrum intravenous antibiotics therapy within 2 weeks prior to initiation of study treatment.
  * Use of any non-study IMP within 3 weeks before initiation of study treatment in this study or ongoing participation in the active treatment phase of another interventional clinical study.
* Have undergone major organ surgery (core needle biopsies are allowed >7 days prior study start), significant trauma, or invasive dental procedures (such as dental implants) within 28 days prior to the initiation of study treatment or plan to undergo elective surgery during the study. Placement of vascular infusion devices is allowed.
* Have received allogeneic hematopoietic stem cell transplantation or organ transplantation.
* Have the following central nervous system metastases:

  * Participants with untreated brain metastases that are symptomatic or large (e.g., >2 cm).
  * Participants who received treatment for central nervous system metastases are not neurologically stable or still on steroids 10 days before initiating IMP of this study.
  * Participants with known leptomeningeal metastases.
* Have active autoimmune disease or history of autoimmune diseases with anticipated relapse (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except for those with clinically stable autoimmune thyroid disease or type 1 diabetes.
* Have had other malignant tumors within 2 years prior to the study treatment are not allowed. Except for those: who have been cured with local treatment (such as basal cell or squamous cell carcinoma of the skin, superficial or non-invasive bladder cancer, carcinoma in situ of the cervix, ductal carcinoma in situ of the breast, papillary carcinoma of thyroid and early stage prostate cancer).
* Have any of the following heart conditions within 6 months prior to the study treatment:

  * Acute coronary syndrome, coronary artery bypass grafting, congestive heart failure, aortic dissection, stroke, or other Grade 3 and above cardiovascular and cerebrovascular events.
  * New York Heart Association functional classification ≥II heart failure or left ventricular ejection fraction <50%.
  * Those who have ventricular arrhythmias requiring clinical intervention, second- to third-degree atrioventricular block, or congenital long QT syndrome. Participants with treated cardiac arrythmia/atrial fibrillation are allowed.
  * Mean QT interval corrected by Fridericia's method >480 ms (the electrocardiogram can be repeated at the discretion of the investigator).
  * Use of cardiac pacemaker.
  * Cardiac troponin I or T >2 x ULN.
* Have any of the following hypertension or diabetic conditions prior to initiation of study treatment:

  * Uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg) while on antihypertensive medicine.
  * Those with a history of hypertensive crisis or hypertensive encephalopathy.
  * Poorly controlled diabetes (fasting blood glucose ≥13.3 mmol/L [240 mg/dL]).
* Have serious non-healing wounds, ulcers, or bone fractures. This includes history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess for which an interval of 6 months must pass before enrollment into this study. In addition, the participant must have undergone correction (or spontaneous healing) of the perforation/fistula and/or the underlying process causing the fistula/perforation.
* Participants with evidence of major coagulation disorders or other significant risks of hemorrhage such as:

  * History of intracranial or intraspinal hemorrhage.
  * Tumor lesions invading large vessels and with significant risk of bleeding
  * Had clinically significant hemoptysis or tumor hemorrhage within 1 month prior to the initiation of study treatment.
* Have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Participants with indwelling catheters (e.g., PleurX) are allowed. However, participants who are clinically stable following treatment for these conditions (including therapeutic thoraco- or paracentesis or with indwelling catheters, e.g., PleurX) are allowed.
* Participants with a history of serious Grade 3 or higher immune-related adverse events (irAEs) that led to treatment discontinuation of a prior immunotherapy. Participants with a history of Grade ≥3 irAEs that did not lead to discontinuation of a prior immunotherapy but fully recovered may be enrolled per investigator's discretion. The investigator may request sponsor guidance in such cases.
* Have a known or suspected hypersensitivity to the study treatments including any active ingredient or excipients thereof.
* Have known human immunodeficiency virus infection or known acquired immunodeficiency syndrome, with the following exceptions:

  * Participants with cluster of differentiation 4 (CD4)+ T-cell (CD4+) counts ≥350 cells/µL per local laboratory should generally be eligible for the study.
  * Participants who have not had an opportunistic infection within the past 12 months.
* Have a known history/positive serology for hepatitis B requiring active antiviral therapy (unless immune due to vaccination or resolved natural infection or unless passive immunization due to immunoglobulin therapy). Individuals with positive serology must have hepatitis B virus viral load below the limit of quantification.
* Have an active hepatitis C virus infection; individuals who have completed curative antiviral treatment with hepatitis C virus viral load below the limit of quantification are allowed.
* Participants with AEs from prior antitumor therapy whose AE(s) have not returned to Grade 1 (graded by NCI CTCAE v5.0 criteria) or below (unless the investigator determines that certain AEs pose no safety risk to participants, such as hair loss, Grade 2 peripheral neuropathy or stable hypothyroidism under hormone replacement therapy) are not eligible for the study.
* Have superior vena cava syndrome or symptoms of spinal cord compression.
* Those with active, or a history of, pneumonitis requiring treatment with steroids, or has active, or a history of, interstitial lung disease. Those with a history of pulmonary fibrosis, or currently diagnosed with severe lung diseases such as interstitial pneumonia, pneumoconiosis, chemical pneumonitis, or any other condition resulting in significant impairment in lung function. Exception: Asymptomatic interstitial changes caused by previous radiation therapy, chemotherapy, or other factors such as smoking are acceptable.
* Have active tuberculosis.
* Have underlying condition(s) that may increase the risk of the combination treatment or complicate the interpretation of AEs, as judged by the investigator, or other scenarios in which the investigator consider the participant as not eligible for the study.
* Are vulnerable individuals, i.e., are individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate. This includes all sponsor, study site, or third party (e.g., contract research organization, vendor) personnel directly involved in the conduct of the sudy and their family members or dependents, as well as all study site personnel otherwise supervised by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment emergent adverse events (TEAEs), adverse events of special interest (AESIs), treatment-related TEAEs, treatment-related serious adverse events (SAEs) and treatment-related treatment emergent SAEs | up to 100 days after the last dose of treatment
  In the combination treatment regimen according to the (US) National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI CTCAE v5.0). By treatment arm and overall.
Occurrence of dose interruption, reduction, and discontinuation of study treatment due to TEAEs | up to 100 days after the last dose of treatment
  By treatment arm and overall.
Objective Response Rate | up to 24 months after completion of study treatment of the last participant
  Defined as the proportion of participants in whom a confirmed complete response (CR) or partial response (PR) (per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1] based on the investigator's assessment) is observed as best overall response. By treatment arm.
Best percentage change from baseline in the tumor size | up to 24 months after completion of study treatment of the last participant
  Based on the investigator's tumor assessment according to RECIST 1.1. Defined as the change from baseline in percent to the minimal tumor size until tumor progression/recurrence or death (whichever comes first). By treatment arm.
Proportion of participants who have achieved early tumor shrinkage | up to 2 months after first dose of treatment
  Defined as ≥10% decrease in the pretreatment sum of diameters at first post-treatment tumor scan in target lesions. By treatment arm.

SECONDARY OUTCOMES:
PK assessment: Maximum concentration (Cmax) derived from serum concentration of investigational medicinal product (IMP) | from pre-dose to 21 days after study treatment
  By treatment arm. Only for the first cycle.
PK assessment: Area under the curve during the dosing interval (AUCtau) values derived from serum concentration of IMP | from pre-dose to 21 days after study treatment
  By treatment arm. Only for the first cycle.
Incidence of detectable BNT327 antidrug antibodies in serum | from pre-dose to 100 days after last dose of study treatment
  By treatment arm and overall.
Duration of Response | up to 24 months after completion of study treatment of the last participant
  Defined as the time from first objective response (CR or PR per RECIST 1.1) to first occurrence of objective tumor progression or death from any cause, whichever occurs first based on investigator's review.
Disease Control Rate | up to 24 months after completion of study treatment of the last participant
  Defined as the proportion of participants in whom a confirmed CR or PR or stable disease (per RECIST 1.1, stable disease assessed at least 6 weeks after first dose) is observed as best overall response based on the investigator's review.
Time to Response | up to 24 months after completion of study treatment of the last participant
  Defined as the time from randomization to first objective response (CR or PR per RECIST 1.1) based on the investigator's review.
Progression-Free Survival (PFS) | up to 24 months after completion of study treatment of the last participant
  Based on the investigator's tumor assessment according to RECIST 1.1. Defined as the time from randomization to first confirmed objective tumor progression (progressive disease per RECIST 1.1), or death from any cause, whichever occurs first.
PFS rate | up to 24 months after completion of study treatment of the last participant
  As measured at 6, 12, 18, and 24 months
Overall Survival (OS) | up to 24 months after completion of study treatment of the last participant
  Defined as the time from randomization to death from any cause
OS rate | up to 24 months after completion of study treatment of the last participant
  As measured at 6, 12, 18, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (64):
- United States (18):
  - Alaska Oncology and Hematology, LLC, Anchorage, Alaska
  - Valkyrie Clinical Trials, Los Angeles, California
  - Clermont Oncology Center, Clermont, Florida
  - Hematology Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Tallahassee Memorial Physician Partners - Cancer & Hematology Specialists, Tallahassee, Florida
  - Carle Foundation Hospital d/b/a Carle Cancer Center, Urbana, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc, Fort Wayne, Indiana
  - University of Kentucky Chandler Medical Center (UKCMC) - Markey Cancer Center (Lucille P. Markey Cancer Center), Lexington, Kentucky
  - Allina Health, Minneapolis, Minnesota
  - SSM Health Cancer Care - St. Clare, Fenton, Missouri
  - Nebraska Hematology-Oncology (NHO) - Lincoln, Lincoln, Nebraska
  - Clinical Research Alliance Inc, Westbury, New York
  - Haywood Infusion Center, Clyde, North Carolina
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - The Christ Hospital Cancer Center, Cincinnati, Ohio
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Millenium Research & Clinical Development, Houston, Texas
  - SSM Health Cancer Care, Madison, Wisconsin
- Australia (5):
  - Lyell McEwin Hospital, Adelaide
  - St. Vincent's Hospital, Fitzroy
  - Peninsula Oncology Centre, Frankston
  - Royal North Shore Hospital, St Leonards
  - Westmead Hospital, Westmead
- South Korea (9):
  - Chungbuk National University Hospital, Cheongju-si
  - Yeungnam University Medical Center, Daegu
  - National Cancer Center, Goyang-si
  - Gachon University Gil Medical Center, Incheon
  - Gyeongsang National University Hospital (GNUH), Jinju
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
  - Ajou University Hospital, Suwon
- Turkey (Türkiye) (21):
  - Baskent University Hospital Adana Dr Turgut Noyan Research Center, Adana
  - Medical Park Seyhan Hospital, Adana
  - Adana City Training and Research Hospital, Adana
  - Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Ankara Etlik Sehir Hastanesi, Ankara
  - Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Hacettepe University Medical Faculty Oncology Hospital, Ankara
  - Memorial Ankara Hospital, Ankara
  - Liv Hospital, Ankara
  - Ankara City Hospital, Ankara
  - Gaziantep Sanko University Medical Faculty, Gaziantep
  - Koc Universitesi Hastanesi (Koc University Hospital), Istanbul
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Acibadem Adana Hastanesi, Istanbul
  - Yeditepe University Kosuyolu Hospital, Istanbul
  - Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Medical Point Izmir Hospital, Izmir
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Sakarya University - Faculty of Medicine, Sakarya
  - Namik Kemal University Hospital, Tekirdağ
  - Gazi University Medical Faculty, Yenimahalle
- United Kingdom (11):
  - Queen Elizabeth Hospital Birmingham - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Velindre Hospital - Velindre NHS Trust, Cardiff
  - Ninewells Hospital and Medical School - Tayside Health Board, Dundee
  - Royal Devon and Exeter Hospital, Wonford - Royal Devon And Exeter NHS Foundation Trust, Exeter
  - Huddersfield Royal Infirmary - Calderdale and Huddersfield NHS Foundation Trust, Huddersfield
  - St James's University Hospital - Leeds Teaching Hospitals NHS Trust, Leeds
  - Sarah Cannon Research Institute, London
  - Northern Centre for Cancer Care,The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Royal Preston Hospital - Lancashire Teaching Hospitals NHS Foundation Trust, Preston
  - Royal Stoke University Hospital - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No